CLINICAL TRIAL: NCT05119114
Title: Role of Volumetric Magnetic Resonance Imaging in Evaluation of Different Types of Dementia
Brief Title: Volumetric Magnetic Resonance Imaging in Dementia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel-Tawab Mohamed, Dr, Assiut University
Other Study IDs: MRI in dementia
Record Dates: First submitted 2021-10-18; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — A standardized multi-parametric MRI protocol will be implemented for all patients. All sequences will be acquired on a 1.5 Tesla scanner. After completion of the MRI study, the digital imaging and communication data will be sent to a diagnostic workstation for post-processing and analysis. Patients of the study will be subjected to detailed structural MRI for detection of signs of neurodegenerative changes. Volumetric high-resolution 3D scans will be used for quantitative study.

SUMMARY:
Dementia is a term for the impaired ability to remember, think, or make decisions that interferes with doing everyday activities. Alzheimer's disease is the most common type of dementia. Though dementia mostly affects older adults, it is not a part of normal aging. This study aims to assess the role of volumetric MRI in evaluation of different types of dementia.

DETAILED DESCRIPTION:
Neurocognitive disorders (dementia) are prevalent clinical problems. With the increase in average life expectancy, its prevalence is rising at an alarming rate. In 2005, an estimated 24 million people around the world suffered from dementia, and that number is expected to double every 20 years. By 2040, it is predicted that over 81 million people worldwide will suffer from dementia. Most experts agree that treatment will be most beneficial if applied early, before significant, potentially irreversible neurodegeneration and functional impairment has occurred.

Clinical symptoms of most subtypes of dementia arise from progressive neuron and synapse loss, with the resulting tissue atrophy. Brain magnetic resonance imaging (MRI) is regularly used in diagnosing dementia as it visualises the structural changes caused by neurodegeneration. It is key in defining subtle differences between healthy and pathological cerebral volume loss and between dementia subtypes.

Visual assessment of brain atrophy patterns is commonly supported through the use of visual rating scales. However, these scales have a subjective element and their application relies heavily on the prior experience of the radiologist using them. And they have poor sensitivity to subtle or prodromal changes and have ceiling and/or floor effects.

Application of quantitative volumetric reporting tools, which automatically quantify an individual patient's regional brain volumes and compare them to healthy populations, can potentially help in interpretation of the severity and distribution of brain atrophy and contextualize their findings by referencing normative brain volumes in healthy populations. This will improve the accuracy of radiological diagnosis of different subtypes of dementia

ELIGIBILITY:
Inclusion Criteria:

* Patients with any type of dementia.
* Patients with mini mental state examination equal or more than 18.

Exclusion Criteria:

* Patients with contra-indications to MRI.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted over the period of 2 years during which all available cases with dementia presented to the Neurology Centre at Assiut university well be investigated.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
MRI Accuracy in dementia | 1 week
  Assess the accuracy of magnetic resonance imaging in differentiate between normal aging and cases of dementia

CONTACTS AND LOCATIONS:
Overall Officials: Hosam A Youssif, MD, Study Director — Assiut University; Ahmed Abdel-Razzak, McS, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ferri CP, Prince M, Brayne C, Brodaty H, Fratiglioni L, Ganguli M, Hall K, Hasegawa K, Hendrie H, Huang Y, Jorm A, Mathers C, Menezes PR, Rimmer E, Scazufca M; Alzheimer's Disease International. Global prevalence of dementia: a Delphi consensus study. Lancet. 2005 Dec 17;366(9503):2112-7. doi: 10.1016/S0140-6736(05)67889-0. PMID 16360788
- [Result] Fennema-Notestine C, Hagler DJ Jr, McEvoy LK, Fleisher AS, Wu EH, Karow DS, Dale AM; Alzheimer's Disease Neuroimaging Initiative. Structural MRI biomarkers for preclinical and mild Alzheimer's disease. Hum Brain Mapp. 2009 Oct;30(10):3238-53. doi: 10.1002/hbm.20744. PMID 19277975
- [Result] Duchesne S, Caroli A, Geroldi C, Barillot C, Frisoni GB, Collins DL. MRI-based automated computer classification of probable AD versus normal controls. IEEE Trans Med Imaging. 2008 Apr;27(4):509-20. doi: 10.1109/TMI.2007.908685. PMID 18390347
- [Result] Ten Kate M, Barkhof F, Boccardi M, Visser PJ, Jack CR Jr, Lovblad KO, Frisoni GB, Scheltens P; Geneva Task Force for the Roadmap of Alzheimer's Biomarkers. Clinical validity of medial temporal atrophy as a biomarker for Alzheimer's disease in the context of a structured 5-phase development framework. Neurobiol Aging. 2017 Apr;52:167-182.e1. doi: 10.1016/j.neurobiolaging.2016.05.024. PMID 28317647